CLINICAL TRIAL: NCT03610711
Title: REACTION (Radiation Enhanced Assessment of Combination Therapies in Immuno-ONcology) - Nivolumab or Nivolumab in Combination With Other Immuno-oncology (IO) Agents After Targeted Systemic Radiation in Patients With Advanced Esophagogastric Cancer
Acronym: REACTION
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: J1884; IRB00166032 (Other: JHM IRB); CA224-053 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Gastroesophageal Cancer; Immune Checkpoint Inhibition
MeSH Terms: interventions — Nivolumab; relatlimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A Nivolumab Only (Experimental): stereotactic body radiation (SBRT) 8G x 3 followed by Nivolumab 240mg administered IV over 30 minutes every 2 weeks for one year or until evidence of disease progression or unresolved toxicity.
  Interventions: Drug: Nivolumab
- Arm B Nivolumab + Relatlimab (Experimental): stereotactic body radiation (SBRT) 8G x 3 followed by Nivolumab 240mg administered IV over 30 minutes every 2 weeks and Relatlimab (anti-LAG3) every 2 weeks for one year or until evidence of disease progression or unresolved toxicity.
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — 240mg administered IV over 30 minutes every 2 weeks for one year
  Other Names: Optivo
Drug: Relatlimab — every 2 weeks for one year
  Other Names: anti-LAG3
  Arms: Arm B Nivolumab + Relatlimab

SUMMARY:
This is a Phase 1B study assessing the safety of immune checkpoint inhibition after SBRT in patients with recurrent or metastatic gastroesophageal cancer (limited metastatic disease).

DETAILED DESCRIPTION:
This is a Phase 1B study assessing the safety of immune checkpoint inhibition after SBRT in patients with recurrent or metastatic gastroesophageal cancer (limited metastatic disease). Arm A explores the safety and efficacy of nivolumab alone, and Arm B explores the safety and efficacy of nivolumab plus Relatlimib. Patients with recurrent or metastatic esophagogastric cancer are eligible for this study which will enroll patients with limited disease burden and who are Programmed death-1(PD-1) therapy naïve. This will allow for us to assess if systemic ablative radiation (SBRT to multiple metastatic sites plus PD-1/ anti-LAG3) is able to enhance the effectiveness of nivolumab +/- anti-LAG3 or to overcome treatment resistance mechanisms. Patients will be treated with targeted high dose radiation (SBRT) to metastatic lesions as outlined below. One of the lesions which is considered the easiest to biopsy and not causing symptoms will not be radiated so as to obtain tissue for correlative analysis. This lesion will then be re-biopsied approx. 4 weeks after the completion of radiation to the other metastatic sites. If a lesion is causing pain or other symptoms this site will not be chosen as the biopsiable site. The chosen metastatic lesion can then be irradiated at a later date if we do not see disease response in that region. Approximately 21 patients will be enrolled on study with 6 enrolled on Arm A, and 15 enrolled on Arm B.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years old.
* Histologically proven (squamous cell or adenocarcinoma) esophageal or gastro-esophageal junction cancer or gastric cancer (core biopsy required)
* Either a formalin fixed paraffin block or a minimum of ten 5-micron tissue section's (slides) of tumor biopsy sample must be available for biomarker evaluation.
* Recurrent disease or Stage IV disease as per American Joint Committee on Cancer (AJCC) staging 8.0 - patients who decline systemic chemotherapy in the first line metastatic setting are eligible.
* (Relatlimab arm only) LVEF assessment with documented left ventricular ejection fraction ( LVEF) >/=50% by either echocardiogram TTE or multigated acquisition scan (MUGA) (TTE preferred test) within 6 months from first study drug administration,whichever is most recent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function as follows:

  * Leukocytes ≥ 2,000/mm3
  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Creatinine ≤ 2.0 mg/dL
  * Bilirubin (total) within normal institutional limits (except subjects with Gilbert Syndrome who must have total bilirubin < 3.0 mg/dL)
  * Aspartate aminotransferase (AST) (SGOT), Alanine Aminotransferase (ALT) (SGPT), and alkaline phosphatase ≤ 2.5 times the institutional upper limit of normal
  * prothrombin time (PT) such that international normalized ratio (INR) is ≤ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) ≤ institutional upper limit of normal
  * Adequate cardiac function as defined by: no evidence of (PR) prolongation or Atrioventricular block (AV block) on baseline electrocardiogram (ECG).
* The effects of nivolumab, relatlimab or BMS-986178, on the developing human fetus are unknown. For this reason women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 5 months after the last dose of nivolumab +/- IO therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Sexually active fertile men must use effective barrier birth control if their partners are WOCBP for 7 months after the last dose of nivolumab +/- IO therapy. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of registration.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (see Appendix 4) for the duration of treatment with study treatment(s) plus 33 weeks after the last dose of the study treatment (ie, 90 days [duration of sperm turnover] plus the time required for nivolumab and relatlimab to undergo approximately 5 half-lives). In addition, male participants must be willing to refrain from sperm donation during this time.
* Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated Institutional Review Board (IRB) approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report Adverse Events (AEs), understand the drug dosing schedule and use of medications to control AEs.

Exclusion Criteria:

* Any active or history of autoimmune disease (including any history of inflammatory bowel disease), or history of syndrome that required systemic steroids or immune-suppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy.
* (Relatlimab arm only) Troponin T (TnT) or I (TnI) > 2 × institutional upper limit of normal (ULN). Subjects with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤1 x ULN. If TnT or TnI levels are > 1 to 2 × ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the BMS Medical Monitor or designee. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the Bristol Myers Squibb (BMS) Medical Monitor or designee.
* (Relatlimab arm only) Participants must not have a history of myocarditis
* (Relatlimab arm only) Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:
* Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
* Uncontrolled angina within the 3 months prior to consent
* Any history of clinically significant arrhythmias (such as ventricular tachycardia, poorly controlled atrial fibrillation, ventricular fibrillation, or torsades de pointes)
* Corrected QT interval (QTc) prolongation > 480 msec
* History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association (NYHA) functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, , poorly controlled venous thrombosis etc.)
* Cardiovascular disease-related requirement for daily supplemental oxygen
* History of two or more MIs OR two or more coronary revascularization procedures
* (Relatlimab arm only) LVEF (Left Ventricular Ejection Fraction) assessment with documented LVEF ≥ 50% by either TTE or MUGA (TTE preferred test) within 6 months from first study drug administration.
* Ongoing requirement for systemic corticosteroids. However, inhalational steroids are allowed.
* Subjects with previous malignancies (except non-melanoma skin cancers, in situ bladder, gastric, breast, colon or cervical cancers/dysplasia) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
* Subjects with known brain metastasis are excluded from this study. Patients with suspected brain metastasis must have brain imaging (either MRI brain or CT brain with contrast) prior to enrollment.
* Subjects with a history of interstitial lung disease. Patients requiring continuous supplemental oxygen are excluded.
* Use of any vaccines against infectious diseases (e.g., influenza, varicella. etc.) within 4 weeks (28 days) of initiation of study therapy.
* Active systemic infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
* Known positive history or positive test for Human Immunodeficiency Virus or Acquired ImmunoDeficiency Syndrome (AIDS).
* History of allergy to study drug components.
* Women who are pregnant or nursing.
* Men with female partners (WOCBP) that are not willing to use contraception
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug or radiation hazardous or obscure the interpretation of toxicity or adverse events.
* Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the infiltrating CD8+ T cell density units after systemic treatment with radiation plus nivolumab +/- Relatlimib | 5 years
  Change in the infiltrating CD8+ T cell density units pre- and post-systemic treatment with radiation plus nivolumab +/- Relatlimib in the non-irradiated metastatic lesion.

SECONDARY OUTCOMES:
Safety profile of nivolumab +/- Relatlimib plus systemic radiation as determined by number of drug-related adverse events | 5 years
  Number of drug-related adverse events Grade 3 or higher as defined by CTCAE 5.0 (CTCAE v5.0).
Efficacy of PD-1 inhibition +/- Relatlimib as determined by number of participants without evidence of disease progression | 3 months post targeted radiation

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lam, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Alleghany Health Network, Pittsburgh, Pennsylvania
  - Baylor University, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of gastric adenocarcinoma. Nature. 2014 Sep 11;513(7517):202-9. doi: 10.1038/nature13480. Epub 2014 Jul 23. PMID 25079317
- [Background] Spranger S, Spaapen RM, Zha Y, Williams J, Meng Y, Ha TT, Gajewski TF. Up-regulation of PD-L1, IDO, and T(regs) in the melanoma tumor microenvironment is driven by CD8(+) T cells. Sci Transl Med. 2013 Aug 28;5(200):200ra116. doi: 10.1126/scitranslmed.3006504. PMID 23986400
- [Background] Thompson ED, Zahurak M, Murphy A, Cornish T, Cuka N, Abdelfatah E, Yang S, Duncan M, Ahuja N, Taube JM, Anders RA, Kelly RJ. Patterns of PD-L1 expression and CD8 T cell infiltration in gastric adenocarcinomas and associated immune stroma. Gut. 2017 May;66(5):794-801. doi: 10.1136/gutjnl-2015-310839. Epub 2016 Jan 22. PMID 26801886
- [Background] Derks S, Nason KS, Liao X, Stachler MD, Liu KX, Liu JB, Sicinska E, Goldberg MS, Freeman GJ, Rodig SJ, Davison JM, Bass AJ. Epithelial PD-L2 Expression Marks Barrett's Esophagus and Esophageal Adenocarcinoma. Cancer Immunol Res. 2015 Oct;3(10):1123-1129. doi: 10.1158/2326-6066.CIR-15-0046. Epub 2015 Jun 16. PMID 26081225
- [Background] Muro K, Chung HC, Shankaran V, Geva R, Catenacci D, Gupta S, Eder JP, Golan T, Le DT, Burtness B, McRee AJ, Lin CC, Pathiraja K, Lunceford J, Emancipator K, Juco J, Koshiji M, Bang YJ. Pembrolizumab for patients with PD-L1-positive advanced gastric cancer (KEYNOTE-012): a multicentre, open-label, phase 1b trial. Lancet Oncol. 2016 Jun;17(6):717-726. doi: 10.1016/S1470-2045(16)00175-3. Epub 2016 May 3. PMID 27157491
- [Background] Derks S, Liao X, Chiaravalli AM, Xu X, Camargo MC, Solcia E, Sessa F, Fleitas T, Freeman GJ, Rodig SJ, Rabkin CS, Bass AJ. Abundant PD-L1 expression in Epstein-Barr Virus-infected gastric cancers. Oncotarget. 2016 May 31;7(22):32925-32. doi: 10.18632/oncotarget.9076. PMID 27147580
- [Background] McGranahan N, Furness AJ, Rosenthal R, Ramskov S, Lyngaa R, Saini SK, Jamal-Hanjani M, Wilson GA, Birkbak NJ, Hiley CT, Watkins TB, Shafi S, Murugaesu N, Mitter R, Akarca AU, Linares J, Marafioti T, Henry JY, Van Allen EM, Miao D, Schilling B, Schadendorf D, Garraway LA, Makarov V, Rizvi NA, Snyder A, Hellmann MD, Merghoub T, Wolchok JD, Shukla SA, Wu CJ, Peggs KS, Chan TA, Hadrup SR, Quezada SA, Swanton C. Clonal neoantigens elicit T cell immunoreactivity and sensitivity to immune checkpoint blockade. Science. 2016 Mar 25;351(6280):1463-9. doi: 10.1126/science.aaf1490. Epub 2016 Mar 3. PMID 26940869
- [Background] Attwood SE, Smyrk TC, DeMeester TR, Mirvish SS, Stein HJ, Hinder RA. Duodenoesophageal reflux and the development of esophageal adenocarcinoma in rats. Surgery. 1992 May;111(5):503-10. PMID 1598670
- [Background] Llosa NJ, Cruise M, Tam A, Wicks EC, Hechenbleikner EM, Taube JM, Blosser RL, Fan H, Wang H, Luber BS, Zhang M, Papadopoulos N, Kinzler KW, Vogelstein B, Sears CL, Anders RA, Pardoll DM, Housseau F. The vigorous immune microenvironment of microsatellite instable colon cancer is balanced by multiple counter-inhibitory checkpoints. Cancer Discov. 2015 Jan;5(1):43-51. doi: 10.1158/2159-8290.CD-14-0863. Epub 2014 Oct 30. PMID 25358689
- [Background] Pera M, Brito MJ, Poulsom R, Riera E, Grande L, Hanby A, Wright NA. Duodenal-content reflux esophagitis induces the development of glandular metaplasia and adenosquamous carcinoma in rats. Carcinogenesis. 2000 Aug;21(8):1587-91. PMID 10910963
- [Background] Zaidi AH, Saldin LT, Kelly LA, Bergal L, Londono R, Kosovec JE, Komatsu Y, Kasi PM, Shetty AA, Keane TJ, Thakkar SJ, Huleihel L, Landreneau RJ, Badylak SF, Jobe BA. MicroRNA signature characterizes primary tumors that metastasize in an esophageal adenocarcinoma rat model. PLoS One. 2015 Mar 31;10(3):e0122375. doi: 10.1371/journal.pone.0122375. eCollection 2015. PMID 25826212
- [Background] Bonde P, Sui G, Dhara S, Wang J, Broor A, Kim IF, Wiley JE, Marti G, Duncan M, Jaffee E, Montgomery E, Maitra A, Harmon JW. Cytogenetic characterization and gene expression profiling in the rat reflux-induced esophageal tumor model. J Thorac Cardiovasc Surg. 2007 Mar;133(3):763-9. doi: 10.1016/j.jtcvs.2006.07.044. PMID 17320581
- [Background] Gibson MK, Zaidi AH, Davison JM, Sanz AF, Hough B, Komatsu Y, Kosovec JE, Bhatt A, Malhotra U, Foxwell T, Rotoloni CL, Hoppo T, Jobe BA. Prevention of Barrett esophagus and esophageal adenocarcinoma by smoothened inhibitor in a rat model of gastroesophageal reflux disease. Ann Surg. 2013 Jul;258(1):82-8. doi: 10.1097/SLA.0b013e318270500d. PMID 23108119
- [Background] Kosovec JE, Zaidi AH, Kelly LA, Rotoloni CL, Vytlacil C, DiCarlo C, Matsui D, Komatsu Y, Boyd NH, Omstead A, Kolano EL, Biederman RW, Finley G, Silverman JF, Landreneau RJ, Jobe BA. Preclinical Study of AUY922, a Novel Hsp90 Inhibitor, in the Treatment of Esophageal Adenocarcinoma. Ann Surg. 2016 Aug;264(2):297-304. doi: 10.1097/SLA.0000000000001467. PMID 26445473
- [Background] Zaidi AH, Kosovec JE, Matsui D, Omstead AN, Raj M, Rao RR, Biederman RWW, Finley GG, Landreneau RJ, Kelly RJ, Jobe BA. PI3K/mTOR Dual Inhibitor, LY3023414, Demonstrates Potent Antitumor Efficacy Against Esophageal Adenocarcinoma in a Rat Model. Ann Surg. 2017 Jul;266(1):91-98. doi: 10.1097/SLA.0000000000001908. PMID 27471841
- [Background] Miyashita T, Shah FA, Marti G, Wang J, Armstrong T, Bonde P, Gibson MK, Yoshimura K, Montgomery EA, Duncan MD, Jaffee EM, Harmon JW. Vaccine impedes the development of reflux-induced esophageal cancer in a surgical rat model: efficacy of the vaccine in a Pre-Barrett's esophagus setting. J Gastrointest Surg. 2008 Jan;12(1):2-7; discussion 7-9. doi: 10.1007/s11605-007-0337-2. Epub 2007 Oct 24. PMID 17957441
- [Background] Kelly RJ, Zaidi AH, Smith MA, Omstead AN, Kosovec JE, Matsui D, Martin SA, DiCarlo C, Werts ED, Silverman JF, Wang DH, Jobe BA. The Dynamic and Transient Immune Microenvironment in Locally Advanced Esophageal Adenocarcinoma Post Chemoradiation. Ann Surg. 2018 Dec;268(6):992-999. doi: 10.1097/SLA.0000000000002410. PMID 28806299
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Finkelstein SE, Timmerman R, McBride WH, Schaue D, Hoffe SE, Mantz CA, Wilson GD. The confluence of stereotactic ablative radiotherapy and tumor immunology. Clin Dev Immunol. 2011;2011:439752. doi: 10.1155/2011/439752. Epub 2011 Nov 15. PMID 22162711
- [Background] Wang X, Schoenhals JE, Li A, Valdecanas DR, Ye H, Zang F, Tang C, Tang M, Liu CG, Liu X, Krishnan S, Allison JP, Sharma P, Hwu P, Komaki R, Overwijk WW, Gomez DR, Chang JY, Hahn SM, Cortez MA, Welsh JW. Suppression of Type I IFN Signaling in Tumors Mediates Resistance to Anti-PD-1 Treatment That Can Be Overcome by Radiotherapy. Cancer Res. 2017 Feb 15;77(4):839-850. doi: 10.1158/0008-5472.CAN-15-3142. Epub 2016 Nov 7. PMID 27821490
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Wong J, Armour E, Kazanzides P, Iordachita I, Tryggestad E, Deng H, Matinfar M, Kennedy C, Liu Z, Chan T, Gray O, Verhaegen F, McNutt T, Ford E, DeWeese TL. High-resolution, small animal radiation research platform with x-ray tomographic guidance capabilities. Int J Radiat Oncol Biol Phys. 2008 Aug 1;71(5):1591-9. doi: 10.1016/j.ijrobp.2008.04.025. PMID 18640502
- [Background] Demaria S, Golden EB, Formenti SC. Role of Local Radiation Therapy in Cancer Immunotherapy. JAMA Oncol. 2015 Dec;1(9):1325-32. doi: 10.1001/jamaoncol.2015.2756. PMID 26270858
- [Background] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Sun J, Dirden-Kramer B, Ito K, Ernst PB, Van Houten N. Antigen-specific T cell activation and proliferation during oral tolerance induction. J Immunol. 1999 May 15;162(10):5868-75. PMID 10229822
- [Background] Carlson CS, Emerson RO, Sherwood AM, Desmarais C, Chung MW, Parsons JM, Steen MS, LaMadrid-Herrmannsfeldt MA, Williamson DW, Livingston RJ, Wu D, Wood BL, Rieder MJ, Robins H. Using synthetic templates to design an unbiased multiplex PCR assay. Nat Commun. 2013;4:2680. doi: 10.1038/ncomms3680. PMID 24157944
- [Background] Robins HS, Campregher PV, Srivastava SK, Wacher A, Turtle CJ, Kahsai O, Riddell SR, Warren EH, Carlson CS. Comprehensive assessment of T-cell receptor beta-chain diversity in alphabeta T cells. Blood. 2009 Nov 5;114(19):4099-107. doi: 10.1182/blood-2009-04-217604. Epub 2009 Aug 25. PMID 19706884
- [Background] Anagnostou V, Smith KN, Forde PM, Niknafs N, Bhattacharya R, White J, Zhang T, Adleff V, Phallen J, Wali N, Hruban C, Guthrie VB, Rodgers K, Naidoo J, Kang H, Sharfman W, Georgiades C, Verde F, Illei P, Li QK, Gabrielson E, Brock MV, Zahnow CA, Baylin SB, Scharpf RB, Brahmer JR, Karchin R, Pardoll DM, Velculescu VE. Evolution of Neoantigen Landscape during Immune Checkpoint Blockade in Non-Small Cell Lung Cancer. Cancer Discov. 2017 Mar;7(3):264-276. doi: 10.1158/2159-8290.CD-16-0828. Epub 2016 Dec 28. PMID 28031159